CLINICAL TRIAL: NCT04568005
Title: Evaluation of Lymphedema Patients Treatment Processes, Health Status, Coronavirus Phobia, Quality of Life, Anxiety and Depression During Covid-19 Pandemic
Brief Title: Evaluation of Lymphedema Patients Status During Covid-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: feyzaakanbegoglu
Record Dates: First submitted 2020-09-25; First posted 2020-09-29 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Lymphedema
Keywords: lymphedema, coronavirus, LYMQOL, HADS
MeSH Terms: conditions — Lymphedema; Coronavirus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The pandemic, which started in China at the end of 2019, appeared in our country in a short time. Most hospitals and physicians were only concerned with the treatment of these patients. One of the most victimized patient groups in this duration was lymphedema patients who were in need of continuous follow-up and rehabilitation at necessary periods, but were also at risk in terms of covid-19 infection and could not go to hospitals unless necessary. The treatment of both primary and secondary lymphedema patients has been interrupted or delayed. This process has affected the health status, treatment processes and quality of life of the lymphedema patient group. The current situation may have caused them anxiety and depression as a result of infection fear. In this study, we aimed to evaluate the treatment processes, health status, coronavirus phobia, anxiety, and depression states of the lymphedema patients .

DETAILED DESCRIPTION:
60 primary and secondary lymphedema male and female patients with stage I,II,III lymphedema older than 18 years old over who were followed up in the lymphedema outpatient clinic of the Physical Medicine and Rehabilitation Clinic were included in the study.They were called by phone. Permission was asked for questioning from the patients reached. A hundred lymphedema patients were called and 60 patients were reached or agreed to be interviewed. The questions on the form and scales were read clearly to the patients who accepted the interview and were asked to be answered by the patient. The health status of the admitted patients during the covid-19 pandemic period and the treatment processes were questioned with the form we prepared.These forms were included socio-demographic features, physical, and detailed medical histories.Edema staging was evaluated by the International Society of Lymphology (ISL) lymphedema staging classification.This information was filled in from patients' files. The pandemic process was evaluated in the other part of the form. Working status, mobilization during the pandemic process, whether he/she or his/her relative was diagnosed with coronavirus infection, whether he/she received suplemental treatment, how much he/she paid attention to hand-foot hygine, whether his/her swelling increased, whether he/she had a cellulite attack, whether he/she regular self-manual lymphatic drainage and/or exercise, It was questioned whether there was an increase in a different symptom other than swelling, eating habits and weight gain, most recently whether he used pressure stocking regularly.In addition, the fear because of the covid-19 virus was questioned with the coronavirus-19 phobia scale (CP19-S), quality of life with lymphedema quality of life arm / leg (LYMQOL), and anxiety and depression with the hospital anxiety and depression scale (HADS).

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary lymphedema patients with stage I,II,II stage
* Aged over 18 years old
* Upper or lower extremity lymphedema

Exclusion Criteria:

* Patients under the age of 18
* Patients who do not accept phone calls.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary or secondary lymphedema patients who aged over 18.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Coronavirus Phobia Scale | 1 day
  The CP19-S has 20 items which is a self-report instrument with a five-point Likert-type scale to assess the levels of coronavirus (covid-19) phobia. All items are rated on a 5 point scale from "strongly disagree (1)" to "strongly agree (5)." The scores on the scale can range between 20 and 100 and a higher score indicates a greater phobia in the respected subscales (psychological, psycho-somatic, economic and social) and total scale. In the present study total scale scores ranged from 20 to 100 .
Lymphedema Quality of Life Arm | 1 day
  The LYMQOL-Arm consists of four domains with 28 items. These domains are symptoms, appearance, function, and mood. The answers were evaluated on a four-point Likert scale (1= not at all 2= a little, 3= quite a bit, 4= a lot). Each item received a score between 1 and 4, with higher scores indicating a worse QOL. Domain totals were calculated by adding the individual scores and dividing the total by the number of questions answered (If >50% of questions per domain were not answered this cannot be calculated *and =0). If the item was not scored and left blank or not applicable, this was scored with a 0. The four domains and their corresponding questions are: Function 1 (a-h), 2,3, Appearance 4,5,6,7,8 Symptoms 9,10,11,12,13,14 and Emotion 15,16,17,18,19,20. Overall QOL (Q21) is scored as the value marked by the patient, between 0-10
Lymphedema Quality of Life Leg | 1 day
  The LYMQOL-Leg consists of 27 items: 26 multiple-choice questions and 1 rating question. It covers four domains: symptoms, appearance, function, and mood. Scoring and calculating is same with the arm scale but differences are; function 1 (a-f), 2,3 appearance 4,5,6,7,8,9,10 symptoms 11,12,13,14,15 and emotion 16,17,18,19,20,21. Overall quality of life (Q22) is scored as the value marked by the patient, between 0-10.
Hospital Anxiety and Depression Scale | 1 day
  It consists of 14 items with two subscales (seven items for anxiety and seven items for depression). Each item is scored 0-3. Each subscale is scored between 0 and 21. The aim of the scale is not to make a diagnosis, but to determine the risk group bt screening anxiety and depression in a short time in patients with physical diseases. The cut-off points of the Turkish version of the HADS were determined as 10 for the anxiety subscale and 7 for the depression subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Feyza Akan Begoğlu, MD, Principal Investigator — Fatih Sultan Mehmet Training and Research Hospital
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No